CLINICAL TRIAL: NCT01881321
Title: Use of Motivational Interviewing to Increase Contraception Use Among Young Women: a Randomized Control Trial
Brief Title: Use of Motivational Interviewing to Increase Contraception Use Among Young Women
Acronym: MI RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 130108
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Unplanned Pregnancy
Keywords: Contraception; Counseling
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Counseling Intervention (Experimental): Contraceptive counseling session based on the principles of motivational interviewing
  Interventions: Behavioral: Counseling Intervention
- Group 2: Usual Care (No Intervention): The standard clinic-based contraceptive counseling with no additional or theory-based contraceptive counseling session

INTERVENTIONS:
Behavioral: Counseling Intervention — 20-40 minute contraceptive counseling session based on the principles of motivational interviewing
  Arms: Group 1: Counseling Intervention

SUMMARY:
Study design: This is a 2-phase study. During the first phase, the investigators developed a contraceptive counseling intervention based on the principles of Motivational Interviewing, trained counselors, and conducted a small pilot study to develop skills and refine the intervention.

The second phase is this feasibility randomized controlled trial (RCT) to compare outcomes between:

Group 1 - Women randomized to a 20-40 minute contraceptive counseling session based on the principles of motivational interviewing, vs.

Group 2 - Women receiving usual clinic care.

Population: Women, aged 15-29 years, presenting to the University of Chicago family planning clinic for termination of an unintended pregnancy.

Hypothesis: A larger proportion of women who are randomized to receive the MI counseling intervention will be using very effective contraception 3 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 15-29 years
2. Presenting for elective termination of an unintended pregnancy
3. Has not had contraceptive counseling from the team.
4. Willing and able to understand and comply with study protocol
5. Willing and able to sign an informed consent in English

Exclusion Criteria:

1. Current pregnancy intended
2. Current pregnancy desired
3. Reason for pregnancy termination not elective (e.g. fetal anomalies, pregnancy resulted from rape or incest)
4. Plans pregnancy within 6 months
5. Has been administered any sedatives or cervical ripening agents
6. For minors, must not be a ward of the state.

Ages: 15 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Use of very effective contraception | up to 3 months after termination of pregnancy appointment

SECONDARY OUTCOMES:
Correct, consistent use of contraceptive method | up to 3 months
Use of any contraceptive method | up to 3 months
Contraceptive method satisfaction | up to 3 months
Intention to continue current method | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Amy Whitaker, MD MS, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Brown BP, Chor J, Hebert LE, Webb ME, Whitaker AK. Shared negative experiences of long-acting reversible contraception and their influence on contraceptive decision-making: a multi-methods study. Contraception. 2019 Apr;99(4):228-232. doi: 10.1016/j.contraception.2019.01.002. Epub 2019 Jan 24. PMID 30685284
- [Derived] Whitaker AK, Quinn MT, Munroe E, Martins SL, Mistretta SQ, Gilliam ML. A motivational interviewing-based counseling intervention to increase postabortion uptake of contraception: A pilot randomized controlled trial. Patient Educ Couns. 2016 Oct;99(10):1663-9. doi: 10.1016/j.pec.2016.05.011. Epub 2016 May 9. PMID 27211225